CLINICAL TRIAL: NCT00038922
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Dose-Escalating, Safety and Exploratory Pharmacogenomic Study of Orally Administered Recombinant Human Interleukin Eleven (rhIL-11) in Patients With Mild to Moderate Left-Sided Ulcerative Colitis
Brief Title: Study Evaluating rhIL-11 in Left-Sided Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Purpose: Treatment
Other Study IDs: 3067K5-114
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2006-05

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Left-Sided; Ulcerative; Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Ulcer; Colitis | interventions — oprelvekin

INTERVENTIONS:
Drug: rhIL-11

SUMMARY:
To explore the safety of orally delivered rhIL-11 in patients with mild to moderate left-sided ulcerative colitis.

To explore the effects of orally administered rhIL-11 on pharmacogenomics in blood samples and in colonic biopsy tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Documented, signed informed consent to participate in this study
* Age greater than or equal to 18 years
* Documented diagnosis of ulcerative colitis by standard clinical criteria, including endoscopy (either flexible sigmoidoscopy or colonoscopy, sufficient to define the proximal limit of disease) with biopsy

Exclusion Criteria:

* Crohn's disease
* Ulcerative proctitis
* Ulcerative colitis extending beyond the splenic flexure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer